CLINICAL TRIAL: NCT05288400
Title: Evaluation of the Clinical Efficacy and Safety of Amlodipine 5mg/ Bisoprolol Fumarate 5mg /Perindopril Arginine 5mg Fixed-dose Combination in Capsule and Free Monotherapy at the Same Dose in Patients With Uncontrolled Essential Hypertension. A Multicentre, Randomized, Open-label, 12-weeks Study.
Brief Title: Evaluation of the Clinical Efficacy and Safety of Amlodipine 5mg/ Bisoprolol Fumarate 5mg /Perindopril Arginine 5mg Fixed-dose Combination in Capsule and Free Monotherapy at the Same Dose in Patients With Uncontrolled Essential Hypertension.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL3-05166-003
Record Dates: First submitted 2022-02-25; First posted 2022-03-21 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Amlodipine; Bisoprolol; Tablets; Perindopril

STUDY DESIGN:
Intervention Model Description: This was a phase III, multicenter, randomized, open-label, controlled study, over a 12-week treatment period with a single-capsule of fixed dose combination (FDC) of Amlodipine 5 mg/ Bisoprolol fumarate 5 mg / Perindopril arginine 5 mg and free monocomponents of Amlodipine 5 mg, Bisoprolol Fumarate 5 mg and Perindopril arginine 5 mg given concomitantly, in 150 patients with uncontrolled essential HT.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): single-capsule of fixed dosed combination (FDC) of amlodipine 5 mg / bisoprolol fumarate 5 mg / perindopril arginine 5 mg
  Interventions: Combination Product: Amlodipine 5mg + bisoprolol fumarate 5mg + perindopril arginine 5mg
- Group B (Active Comparator): Free triple therapy of amlodipine 5 mg + bisoprolol fumarate 5 mg + perindopril arginine 5 mg, given concomitantly
  Interventions: Drug: Norvasc 5mg tablet; Drug: Concor 5mg tablet; Drug: Coversyl 5mg tablet

INTERVENTIONS:
Combination Product: Amlodipine 5mg + bisoprolol fumarate 5mg + perindopril arginine 5mg — 1 capsule/day Oral administration
  Arms: Group A
Drug: Norvasc 5mg tablet — Norvasc (amlodipine) 5mg, 1 tablet/day
  Arms: Group B
Drug: Concor 5mg tablet — Concor (bisoprolol fumarate) 5mg, 1 tablet/day
  Arms: Group B
Drug: Coversyl 5mg tablet — Coversyl (perindopril arginine) 5mg, 1 tablet/day
  Arms: Group B

SUMMARY:
The purpose of this study was to evaluate the efficacy and the safety of a fixed-dose combination in capsule of Amlodipine 5mg/ Bisoprolol fumarate 5mg/ Perindopril arginine 5mg, and free monotherapy at the same dose in patients with uncontrolled essential hypertension.

DETAILED DESCRIPTION:
This was a phase III, multicenter, randomized, open-label, controlled study, over a 12-week treatment period with a single-capsule of fixed dose combination (FDC) of Amlodipine 5 mg/ Bisoprolol fumarate 5 mg / Perindopril arginine 5 mg and free monocomponents of Amlodipine 5 mg, Bisoprolol fumarate 5 mg and Perindopril arginine 5 mg given concomitantly, in 150 patients with uncontrolled essential HT.

Patients without any non-selection criteria, already treated by anti-hypertensive monotherapy at maximal dose or either by a dual therapy at minimum dose, other than study treatment, having an uncontrolled HT defined by SBP (Systolic Blood Pressure) ≥ 140 and <160 mmHg and DBP (Diastolic Blood Pressure) ≥ 90 and <100 mmHg (in supine position) at 2 different visits (selection and inclusion) were to be selected in this study and randomized to one of two treatment groups: single-capsule combination or free therapy without any wash-out period.

For all patients, controlled blood pressure (BP) was defined as SBP < 140 mmHg and DBP < 90 mmHg.

ELIGIBILITY:
Selection criteria:

* Men or women of any ethnic origin ≥18 years old who signed Informed consent form.
* Patients with uncontrolled hypertension defined by SBP ≥140 and < 160 mmHg and DBP ≥90 and < 100 mmHg already treated by anti-hypertensive monotherapy at maximal dose or either by a dual therapy at minimum dose, other than study treatment (amlodipine or bisoprolol or perindopril), for at least 4 weeks.
* Women of potential childbearing and men (and/or their partners) must agree to use appropriate contraceptive measures. This applies since signing of the Informed Consent form until the last study drug administration.
* Willing to provide signed and dated informed consent.

Non selection criteria

* Unlikely to co-operate in the study, to comply with study treatment or with the study visits.
* Pregnancy, breastfeeding.
* Current participation in another randomized study or within the preceding 3 months.
* Participant already enrolled in the study.
* Alcohol or drug abuse and/or dependence.
* Body mass index > 32 kg/m².
* Grapefruit juice was forbidden during the study (interaction with amlodipine).

Concerning Hypertension (HT)

* DBP ≥100 mmHg and/or SBP ≥160 mmHg under treatment.
* Known or suspected symptomatic orthostatic hypotension.
* HT known to be resistant to Calcium Channel Blockers or Angiotensin Converting Enzyme (ACE) inhibitors or Beta Blockers.
* Secondary HT.
* Complicated HT: known stage III or IV hypertensive retinopathy, macroalbuminuria (patients with microalbuminuria could be selected).

Concerning concomitant diseases

* History of renal disease: Known renal impairment: Patients having a creatinine clearance value classifying them as moderate or severe renal failure (using national or international classification of chronic kidney disease), whatever the method for calculation used (Modification of Diet in Renal Disease (MDRD) or Cockcroft or any other Estimated Glomerular Filtration Rate (eGFR) formula), or bilateral renal artery stenosis or stenosis to a solitary kidney.
* History of cerebrovascular disease: ischemic stroke, cerebral hemorrhage, transient ischemic attack.
* History of heart disease: shock (including cardiogenic), myocardial infarction (within previous 6 months before selection), heart failure class II to IV NYHA (New York Heart Association), coronary revascularization (within the previous 6 months), severe aortic or mitral valve stenosis or hypertrophic obstructive myocardiopathy, unstable angina pectoris (including Prinzmetal's angina).
* History of recent (within previous 6 months before selection, accordingly to the doctor decision) ventricular rhythm disorders (except isolated extrasystoles), atrial fibrillation or atrial flutter, second or third degree atrioventricular (AV) block or other cardiac rhythm disorders leading to important beat-to-beat variations in BP (Left Ventricular Hypertrophy was authorized at selection and during the study).
* Known prolonged QT interval.
* Patients having resting HR <50 bpm.
* History of sick sinus syndrome.
* History of bradycardia clinically significant episode.
* Severe forms of peripheral arterial occlusive disease or severe forms of Raynaud's syndrome.
* Severe bronchial asthma or severe chronic obstructive pulmonary disease.
* Severe gastro-intestinal tract disorders with possible influence on drug absorption or electrolytes.
* Known complicated liver disease (for example: chronic hepatitis, cirrhosis, hepatic encephalopathy…).
* Chronic pancreatitis.
* Endocrine diseases: uncontrolled dysthyroidia, Cushing's syndrome, acromegalia, hyperparathyroidia.
* Diabetes mellitus type I and type II under treatment (patients with diabetes type II well controlled at the selection visit by lifestyle and dietary rules alone could be selected).
* Any history or known severe disease likely to interfere with the conduct of the study, severe evolutive infection, evolutive malignant neoplasm.
* History of neutropenia.
* History of connective tissue disorders (systemic lupus erythematosus, progressive systemic sclerosis or other connective tissue disorders).
* History of severe mental or psychiatric disorder, severe depression or history of severe depression, e.g. requiring hospitalization or at high risk of suicide attempt.
* History of angioneurotic oedema.

Concerning concomitant medications

* β-blockers even if used for other reason than HT, in order to avoid the AE related to the immediate switch during selection visit.
* Antihypertensive treatments having central mechanism of action in order to avoid possible rebound effect at a full immediate stop at the randomization.
* Antiarrhythmic treatments in order to avoid possible interactions with bisoprolol.
* Inability to stop any of the medications listed in the prohibited concomitant medication list.
* Potassium supplement at selection and inclusion visit.
* Drugs contraindicated with the study treatments as defined in the Summaries of Product Characteristics of each study drugs

Concerning contra-indications to treatment with amlodipine, bisoprolol or perindopril

* Any history of angioedema, hereditary, idiopathic or associated with previous ACE inhibitor therapy.
* Allergy / hypersensitivity / history of intolerance or any contra-indications related to:

  * amlodipine or any other dihydropyridine and calcium inhibitors;
  * perindopril or any other ACE inhibitor;
  * bisoprolol or other beta-blockers;
  * any of the excipients of the study drugs.

Inclusion criteria :

* Respect of the previous selection and non-selection criteria.
* Confirmed essential uncontrolled HT under patient's current treatment at W000 visit, defined as SBP ≥140 and < 160 mmHg and DBP ≥90 and < 100 mmHg, measured with a validated automatic device in supine position after at least 10 minutes of rest. There were 3 BP measurements at 2-3 minutes of an interval between each measurement. The mean of the two last values of the three measurements was taken.
* Normal or without any clinically significant abnormality 12-lead ECG (left ventricular hypertrophy and post-MI ECG-changes are authorized at selection and during the study).
* Normal or without clinically significant abnormality of laboratory examinations. Microalbuminuria was authorized.

Non-inclusion criteria :

* As per non-selection criteria.
* Occurrence of an event requiring immediate notification since Selection.
* Laboratory results unavailable at the inclusion visit.
* Withdrawal of informed consent by patient.
* DBP ≥100 mmHg and/or SBP ≥160 mmHg under treatment since the selection visit.
* Positive orthostatic test at inclusion.
* Positive β-human Chorionic Gonadotrophin (β-HCG) pregnancy test (Blood test).
* Laboratory results unavailable at the inclusion visit or clinically significant abnormalities. Macroalbuminuria (>300 mg albumin/24h) was not authorized. ASpartate (Amino)Transferase (ASAT) or ALanine (Amino)Transferase (ALAT) ≥ 2 UNL (Upper Normal Limit) was not authorized.

If all Inclusion and non-inclusion criteria were satisfied, the patient was included and randomized to a treatment group.

Exclusion Criteria (withdrawal criteria) :

* Patients whose BP was still uncontrolled at two consecutive visits (SBP ≥ 140 mmHg or DBP ≥ 90 mmHg) or whose SBP/DBP was above 160/100 mmHg (confirmed with 2 consecutive visits starting W004, at least 14 days apart).
* Onset of an adverse event (AE) which required prescription of a treatment incompatible with the protocol.
* Onset of an AE which, according to the investigator, makes it unsafe for the patient to continue with the study treatment. This includes clinically significant abnormal biochemical and haematological parameters, or clinically significant ECG abnormality.
* Pregnancy.
* Major protocol deviation preventing the analysis of the main endpoint, or which, in the opinion of the investigator, makes it unsafe for the patient to continue to take the study medication and to stay in the study.
* Non-medical reason (patient's personal decision to stop treatment).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline of blood pressure (SBP and DBP) | at baseline, 4, 8 and 12 weeks

SECONDARY OUTCOMES:
Blood pressure control rate (SBP < 140 mmHg and DBP < 90 mmHg) | at 4, 8 and 12 weeks
Response rate for antihypertensive therapy | at 4, 8 and 12 weeks
  Rate of patients with supine blood pressure normalized (SBP <140 mmHg and DBP <90 mmHg) or decrease of SBP ≥20 mmHg and/or decrease of DBP ≥10 mmHg from baseline
Assessment of patient treatment satisfaction TSQM-9 questionnaire | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Konradi, Principal Investigator — Almazov National Medical Research Centre - Department of Hypertension, Saint Petersburg, Russia
Locations (15):
- Russia (15):
  - Regional state budget health care institution "Altai Regional Cardiological dispensary" 46 Malakhova St., Barnaul, Altayskiy Kray
  - Problems of Cardiovascular Diseases" 6 Sosnovy Bulvar St., Kemerovo
  - Autonomous non-profit organization "Medical Center "Alliance" 12 Molodezhnaya St., 12, Kirovsk
  - State budgetary healthcare institution of city of Moscow "City polyclinic #2 of Healthcare Department of city of Moscow" 12 Fruktovaya St., Moscow
  - Federal State Budgetary Institution ''Ourpatient clinic #5'' of the Administration of the President of the Russian Federation 14 Plyushchikha St., Moscow
  - St. Petersburg State Budgetary Healthcare Institution "The city hospital No.38. named after N.A. Semashko" 7/2 letter A Gospitalnaya Str., Pushkin, Saint Pertersburg
  - Pavlov First Saint Petersburg State Medical University L'va Tolstogo str. 6-8, Saint Pertersburg
  - LLC "Medicinskie tekhnologii", Nevzorova street, 6/191025, Saint-Petersburg, Vosstania street, 8 lit A, Saint Petersburg
  - LLC "Strategicheskie Medicinskie Sistemy", Nevzorova street, 6, Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "City outpatient clinic №109" 8 bld. 2 Oleko Dundicha, Saint Petersburg
  - Limited Liability Company "Medical Research Institute" 25 Let. A 3 Kolya Tomchak St., Saint Petersburg
  - Federal State Budgetary Institution "North-West Federal Medical Research Center n.a. V.A. Almazov" of the Ministry of Health of the Russian Federation 2 Akkuratova St., Saint Petersburg
  - The Federal State Budgetary Institute "The Nikiforov Russian Center of Emergency and Radiation Medicine" The Ministry of Russian Federation for Civil Defense, Emergencies and Elimination of Consequences of Natural Disasters, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Consulting and Diagnostic Center No. 85" 89 bld. 3 Let. A Prospekt Veteranov, Saint Petersburg
  - Limited Liability Company "MART" 54 bld. 3 Let. J Maly Prospekt V.O, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/